CLINICAL TRIAL: NCT06962995
Title: Multi-Cancer Detection Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-000321; NCI-2025-03276 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection; Specimen Handling; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Securely stored, de-identified samples and information will be used for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete surveys and have their medical records reviewed on study. Patients may undergo blood or buccal swab and urine sample collection on study.
  Interventions: Procedure: Blood Sample; Other: Surveys

INTERVENTIONS:
Procedure: Blood Sample — Up to 60 mL (about 4-5 Tbsp) of blood may be collected for an initial blood draw and up to 30 mL (about 2-3 Tbsp) may be collected for a second blood draw, 25-45 days after first blood draw. The research blood will be collected at the time of a clinical blood draw, if possible.
  Other Names: Biological Sample Collection; Biospecimen Collection; Specimen Collection; Blood Sample Collection
Other: Surveys — Participants will complete surveys related to attitudes and beliefs around Multi-Cancer Detection testing.

SUMMARY:
This study assesses the incorporation of Multi-Cancer Detection (MCD) testing, designed to detect many types of cancer, into clinical practice to understand both its use and effect in real world practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Has Mayo Clinic medical record number
* Has undergone (within last 6 months) or scheduled to undergo a multi-cancer detection test (MCD) as ordered by provider
* Able to provide informed consent
* ≥ 21 years old
* Ability to provide blood sample

Exclusion Criteria:

* Individuals who have situations that would limit compliance with the study requirements
* Institutionalized (i.e. Federal Medical Prison)
* Known pregnancy (self-reported)
* Currently undergoing active cancer treatment other than adjuvant hormone therapy
* Invasive cancer diagnosis within the last 3 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants who have undergone multi-cancer detection testing (MCD) as part of their clinical care at or outside Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Financial impact of MCD testing | Up to 5 years
  Assessed by types of diagnostic studies ordered as a result of positive MCD test results (e.g., to establish or rule out a cancer diagnosis).
Positive actionable MCD results | Up to 5 years
  Assessed by the number of participants who receive positive MCD results
Psychological Impact of MCD Testing | Baseline (after receiving MCD results)
  Assessed with the Multidimensional Impact of Cancer Risk Assessment (Adapted MICRA), which asks participants to evaluate their response to MCD test results over the past week. The MICRA consists of 20 items answered on a 4-point scale (Never, Rarely, Sometimes, Often). Higher scores generally indicate higher levels of distress or psychological impact.
Change in Patient Satisfaction with MCD Test | Baseline; After receiving MCD results (up to 5 years)
  Participants will complete a 3-question survey, "Satisfaction with the Multi-Cancer Detection Test." Items are answered on a 5-point scale (not at all, a little, somewhat, very, extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Jewel Samadder, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials